CLINICAL TRIAL: NCT01889706
Title: Application of Metformin as Adjuvant Therapy in Overweight and Obese Patients With Type 1 Diabetes Mellitus.
Brief Title: Metformin Therapy in Type 1 Diabetes Mellitus.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Poznan University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Agnieszka Zawada, MD, Poznan University of Medical Sciences
Other Study IDs: MTiT1DM
Record Dates: First submitted 2013-06-25; First posted 2013-06-28 (Estimated); Last update posted 2013-06-28 (Estimated); Status verified 2013-06

CONDITIONS: Loss of Control of Diabetes
Keywords: Type 1 diabetes mellitus,; metformin,; insulin resistance,; obesity
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Insulin Resistance; Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The use of exogenous insulin and incorrect nutritional habits are conducive to obesity and excess weight. This leads to the development of insulin resistance, even in patients with type 1 diabetes mellitus. The purpose of this study is to assess the effects of metformin as adjunctive therapy on anthropometric parameters, insulin resistance and metabolic control in overweight and obese patients with type 1 diabetes mellitus.

The study group consists of 200 Caucasian type 1 diabetic patients with elevated adipose tissue content as measured by electrical bioimpedance, treated at the Poznan University of Medical Sciences Department of Diabetology in 2009-2014. All patients have type 1 diabetes diagnosed by autoimmune antibodies, and are treated with intensive insulin therapy. This group is divided into metformin treated arm (group I+ M, 100 subjects), the remaining 100 patients are treated with insulin alone (control group, group I). Metformin is administered at least 6 months at a mean dose of 1000 mg/day.

The investigators would like to assess the impact of metformin treatment on metabolic control, insulin resistance and anthropometric parameters in overweight and obese patients with type 1 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years <60 years,
* duration of diabetes >3 years,
* lack of metabolic control- HbA1C>7,5% (despite participation in 5-day WHO education program)
* treated with intensive insulin therapy

Exclusion Criteria:

* metabolically decompensate diabetes with acetonuria,
* suspected lack of compliance,
* lack of glucose and ketones self-monitoring,
* hypoglycaemic unawareness or recurrent severe hypoglycemia (defined as more than two episodes of hypoglycemia lowered than 60 mg/dl with loss of consciousness, required assistance to treat) in the past 3 months,
* recurrent diabetic ketoacidosis (more than two episodes in the past year)
* another serious medical illness,
* pregnancy or sexually active woman unwilling to take birth control.
* renal impairment (estimated on the value calculated glomerular filtration rate using the MDRD formula-estimated glomerular filtration rate, eGFR<45 mL / min
* liver cell damage Alanine aminotransferase (ALT), Aspartate aminotransferase (AST) greater than twice the upper normal limit),
* history of drug or alcohol abuse or those who used this drug before
* changes in the way of antihypertensive and antihyperlipemic treatment.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: 200 Caucasian patients with type 1 diabetes admitted to the Department of Internal Medicine and Diabetology, Poznan University of Medical Sciences in years 2009-2014, treated with intensive insulintherapy.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2009-01; Primary Completion 2013-03 (Actual); Study Completion 2014-02 (Estimated)

PRIMARY OUTCOMES:
Body fat content and anthropometric parameters | 6 months
  assessed by electrical bioimpedance using a Tanita BC-418 MA device,

SECONDARY OUTCOMES:
Assessment of metabolic control | 6 months
  (HbA1C, lipid profile)
Insulin requirement | 3 , 6 months

OTHER OUTCOMES:
Assessment of skin AGE | 6 months
  AGE-Reader ( Diagn-Optic)

CONTACTS AND LOCATIONS:
Overall Officials: Dariusz Naskręt, PhD, Principal Investigator — Poznań University of Medical Sciences
Locations (1):
- Department of Internal Medicine and Diabetology, Raszeja Hospital, Poznan, Great Poland, Poland